CLINICAL TRIAL: NCT04049513
Title: A Phase I Dose Escalation Trial of Autologous Third-generation Anti-CD19 Chimeric Antigen Receptor T-cells (WZTL-002) for Relapsed and Refractory B-cell Lymphomas
Brief Title: ENABLE-1 (Engaging Toll-like Receptor Signalling for B-cell Lymphoma Chimeric Antigen Receptor Therapy)
Acronym: ENABLE-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Malaghan Institute of Medical Research (Other)
Collaborators: Wellington Zhaotai Therapies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WZTL002-1; U1111-1216-2053 (Other: World Health Organisation)
Record Dates: First submitted 2019-07-29; First posted 2019-08-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell; Diffuse Large B-cell Lymphoma (DLBCL); Primary Mediastinal B-cell Lymphoma (PMBCL); Transformed Follicular Lymphoma (TFL); Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL)
Keywords: Lymphomas Non-Hodgkin's B-Cell; Chimeric antigen receptor T-cell
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Modified 3+3 dose escalation scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WZTL002-1 (1928T2z CAR T-cells) (Experimental): A starting WZTL-002 dose of 5 × 10^4 CAR T-cells/kg has been selected with four possible dose level cohorts proposed.
  Escalation to a higher dose cohort will be based on assessment of dose limiting toxicities to determine safety at a given dose level.
  Interventions: Biological: WZTL002-1 (1928T2z CAR-T cells); Drug: Cyclophosphamide and Fludarabine lymphodepleting chemotherapy

INTERVENTIONS:
Biological: WZTL002-1 (1928T2z CAR-T cells) — WZTL-002 comprises autologous third-generation anti-CD19 chimeric antigen receptor T-cells (termed 1928T2z). The chimeric antigen receptor in WZTL-002 incorporates the FMC63 anti-CD19 soluble chain variable fragment extracellularly, and portions of both CD28 and the Toll/interleukin-1 receptor (TIR) domain of Toll Like Receptor 2 (TLR2) as intracellular co-stimulatory domains, alongside CD3ζ. WZTL-002 (autologous 1928T2z CAR T-cells) will be administered on D0 as a single IV infusion, following lymphodepleting chemotherapy.
Drug: Cyclophosphamide and Fludarabine lymphodepleting chemotherapy — Cyclophosphamide 500 mg/m^2 IV on days -5 to -3, inclusive. Fludarabine 30 mg/m^2 IV on days -5 to -3, inclusive

SUMMARY:
This Phase 1, single centre, open label dose escalation study aims to identify a safe dose of third-generation anti-CD19 CAR T-cells (WZTL-002) in the treatment of patients with relapsed or refractory (r/r) B-cell Non Hodgkin Lymphoma, for use in further efficacy trials. An expansion cohort will assess automated closed-system manufacture of WZTL-002 and outpatient management of participants.

DETAILED DESCRIPTION:
This is a Phase 1 study, designed to evaluate the safety, feasibility, efficacy and kinetics of third-generation autologous anti-CD19 CAR T-cells, WZTL-002, in patients with relapsed or refractory B-cell Non-Hodgkin Lymphoma without other curative options. The initial dose escalation cohort will use a 3+3 dose escalation design to identify a Maximum Tolerated Dose (MTD) of WZTL-002 using pre-defined Dose Limiting Toxicity (DLT) criteria. Within a subsequent dose expansion cohort at the recommended phase 2 dose, an automated closed-system manufacturing process for WZTL-002 and outpatient clinical management will be implemented.

Eligible participants will undergo leukapheresis to harvest peripheral blood mononuclear cells, the starting material for the manufacture of the autologous third generation anti-CD19 CAR T-cell product, WZTL-002. After WZTL-002 manufacture and confirmation that product release criteria are met, participants will receive lymphodepleting chemotherapy comprising fludarabine and cyclophosphamide on days -5 to day -3, inclusive. WZTL-002 will be administered intravenously on day 0 as a single dose.

Following WZTL-002 administration, participants will be monitored closely for 14 days, including targeted assessments for the specific CAR T-cell related toxicities of Cytokine Release Syndrome (CRS) and Immune Effector Cell Neurotoxicity Syndrome (ICANS). Initial DLT assessment will occur at day 21 after WZTL-002 infusion. A PET/CT Scan to assess treatment response will take place 3 months after WZTL-002 infusion, marking the end of the primary follow up period. The secondary follow up period will occur between 3 months up until 2 years after WZTL-002 treatment. Long term follow up within the trial will occur annually from 2 to 5 years after WZTL-002 treatment, with further follow-up within the Center for International Blood and Marrow Transplant Research (CIBMT) Cellular Therapies Registry and the Australasian Bone Marrow Transplant Recipient Registry (ABMTRR). In addition to clinical data, this study incorporates sample collection for exploratory endpoints including serum cytokine profile following WZTL-002 infusion, and WZTL-002 expansion, persistence and phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to 75 years (inclusive)
* Biopsy-proven relapsed or treatment refractory aggressive B-cell non-Hodgkin lymphoma of the following subtypes per World Health Organisation (WHO) classification: DLBCL and its variants, PMBCL, tFL, FL, MCL
* Requirement for treatment in the opinion of the investigator
* Presence of measurable disease as per Lugano 2014 Criteria
* No other curative treatments available, or not suitable due to patient or disease characteristics or lack of stem cell donor
* Malignancy documented to express CD19 based on flow cytometric or immunohistochemical staining
* Provision of written informed consent for this study
* Lymphoma-related life expectancy at least 12 weeks, and life-expectancy from non-lymphoma related causes of > 12 months
* European Cooperative Oncology Group (ECOG) performance status of 0 to 2 inclusive
* Adequate haematologic function, defined by neutrophils ≥ 1.0 × 10^9/L and platelets ≥ 50 × 10^9/L
* No serious cardiac, pulmonary, hepatic or renal disease.

  * Serum bilirubin < 2.5 times Upper limit of normal (ULN)
  * Estimated creatinine clearance (CrCl) ≥ 50 mL/min using the modified Cockroft Gault estimation or as assessed by direct measurement
  * Cardiac Ejection Fraction ≥ 50% as determined by Echocardiogram or MUGA Scan
  * Oxygen saturations > 92% on room air
  * Diffuse Capacity of the lungs for carbon monoxide (DLCO) or Carbon monoxide transfer coefficient (KCO), Forced expiratory volume in one second (FEV1) and Forced Vital Capacity (FVC) are all ≥ 50% of predicted by spirometry after correcting for haemoglobin and/or volume on lung function testing.

Exclusion Criteria:

* Confirmed active or prior central nervous system (CNS) involvement by lymphoma. In patients with a clinical suspicion of CNS disease, lumbar puncture and MRI brain must be performed
* Active CNS pathology including: epilepsy, seizure within the preceding year, aphasia, paresis, stroke, dementia, psychosis within the preceding year, severe brain injury, Parkinson disease, or cerebellar disease
* Richter Syndrome
* Active autoimmune disease requiring systemic immunosuppression
* Prior solid organ transplantation
* Allogeneic stem cell transplantation within the preceding three months or still requiring systemic immunosuppression
* Current grade II - IV acute graft versus host disease (GVHD), any prior grade IV acute GVHD, or current moderate or severe chronic GVHD
* Systemic corticosteroids at doses of ≥ 20mg prednisone daily or equivalent within 7 days of enrolment
* Peripheral blood lymphocytes < 0.3 x 10^9/L as assessed by complete blood count
* Peripheral blood CD3+ T cells < 150/μL as assessed by lymphocyte subset analysis
* Pregnant or lactating female
* Women of child-bearing potential who are not willing to use highly effective methods of contraception during study participation and for at least 1 year after WZTL-002 administration
* Men who are not willing to use highly effective methods of contraception during study participation and for at least 1 year after WZTL-002 administration
* Men who have a pregnant partner and are not willing to use a condom while performing sexual activity during study participation and for at least 3 months after WZTL-002 administration
* Participants with known sensitivity to immunoglobulin or to components of the investigational product (IP)
* History of active malignancy other than B-cell malignancy within two years prior to enrolment, with the exception of: adequately treated in situ carcinoma of the cervix; adequately treated basal cell carcinoma (BCC) or localized squamous cell carcinoma (SCC) of the skin; other localised malignancy surgically resected (or radically treated with another treatment modality) with curative intent
* Current or prior human immunodeficiency virus (HIV) infection
* Vaccination with a live virus within the preceding four weeks
* Treatment with a purine analogue within the preceding four weeks
* Treatment with alemtuzumab within the preceding 12 weeks
* Cytotoxic chemotherapy, radiotherapy or monoclonal antibody therapy (other than alemtuzumab) within 2 weeks of enrolment
* Prior gene therapy, including prior anti-CD19 chimeric antigen receptor T-cell therapy
* Receipt of an investigational medicine within another clinical trial within the preceding four weeks
* Inadequately controlled systemic infection
* Serologic status reflecting active viral hepatitis B or any history of hepatitis C infection as follows:

  * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU), and if they are willing to receive appropriate anti-viral prophylaxis.
  * Presence of hepatitis C virus (HCV) antibody
* Presence of New York Heart Association (NYHA) class 2 or higher cardiac symptoms not related to lymphoma
* Significant concomitant illnesses which would in the investigator's opinion make the patient an unsuitable candidate for the trial
* Participants who have diminished capacity or any circumstance that would prohibit them from understanding and providing informed consent in accordance with ICH-GCP (International Conference on Harmonisation, Good Clinical Practice)
* Participant does not provide consent to enrol onto International Cellular Therapy Registry

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number and severity of adverse events assessed by CTCAE v5.0, except for Cytokine Release Syndrome and Immune Effector Cell-Associated Neurotoxicity Syndrome, which will be assessed by ASTCT consensus grading criteria | 3 months after administration
  Determine the safety profile of WZTL-002, anti-CD19 CAR T-cells by measuring frequency and severity of adverse events

SECONDARY OUTCOMES:
Feasibility of Manufacture | 3 months after administration
  To investigate the feasibility of manufacture and treatment with WZTL-002, as determined by the proportion of enrolled participants undergoing at least one study leukapheresis procedure that receive WZTL-002
Overall Response Rate | 3 months after administration
  To estimate the overall response rate (ORR) as determined by complete response (CR) plus partial response (PR) 3 months after WZTL-002 administration
Cumulative CR rate | 6 months after administration
  To determine the cumulative CR rate 6 months after WZTL-002 administration
Relapse-free survival | 24 months after administration
  To estimate the relapse-free survival (RFS) for subjects treated with WZTL-002 over a period of 24 months after WZTL-002 administration
Overall survival | 24 months after administration
  To estimate the overall survival (OS) distribution for subjects treated with WZTL-002 over a period of 24 months after WZTL-002 administration
Recommended dose | 3 months after administration
  To determine the recommended phase 2 dose of WZTL-002 for treatment of R/R B-NHL

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weinkove, MBBS, PhD, Principal Investigator — Te Whatu Ora Health New Zealand Capital Coast & Hutt Valley
Locations (1):
- Wellington Hospital, Te Whatu Ora Health New Zealand Capital Coast & Hutt Valley, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication

REFERENCES:
- [Background] George P, Dasyam N, Giunti G, Mester B, Bauer E, Andrews B, Perera T, Ostapowicz T, Frampton C, Li P, Ritchie D, Bollard CM, Hermans IF, Weinkove R. Third-generation anti-CD19 chimeric antigen receptor T-cells incorporating a TLR2 domain for relapsed or refractory B-cell lymphoma: a phase I clinical trial protocol (ENABLE). BMJ Open. 2020 Feb 9;10(2):e034629. doi: 10.1136/bmjopen-2019-034629. PMID 32041862
- [Derived] Weinkove R, George P, Ruka M, Haira TH, Giunti G. Chimeric antigen receptor T-cells in New Zealand: challenges and opportunities. N Z Med J. 2021 Sep 17;134(1542):96-108. PMID 34531588
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Dasyam N, George P, Weinkove R. Chimeric antigen receptor T-cell therapies: Optimising the dose. Br J Clin Pharmacol. 2020 Sep;86(9):1678-1689. doi: 10.1111/bcp.14281. Epub 2020 Mar 24. PMID 32175617